CLINICAL TRIAL: NCT04401592
Title: The Role of Galectin-1,3,9 in the the Non-invasive Diagnosis of Endometriosis
Brief Title: The Role of Galectins in the Non-invasive Diagnosis of Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Semmelweis University (Other)
Collaborators: University of Pecs (Other)
Responsible Party: Principal Investigator, Reka Brubel, MD PhD, Semmelweis University
Other Study IDs: ENDOGAL
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-05

CONDITIONS: Endometriosis; Endometriosis Ovary; Endometriosis Rectovaginal Septum
Keywords: Endometriosis; Biomarker; Non-invasive diagnosis; Galectins
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- disease and control

SUMMARY:
Endometriosis is one of the most common infertility-related gynecologic disorder that affect approximately 10-15% of women in reproductive age. The main symptoms are chronic pelvic pain, infertility, dysmenorrhea and dyspareunia. There exists an average diagnostic delay of 7 year but data widely varies between different countries. The current "gold standard" in the diagnosis of endometriosis remains a laparoscopy. Since laparoscopy is an invasive surgical procedure with its potential risk, the development of a non-invasive laboratory test would be of great benefit in the early, clinical management of this diseaseIn the past few years, lectins have become the focus of reproductive immunology, inflammation and autoimmunity. Galectins (Gal) are beta-galactoside binding lectins that play a key role in the regulation of the immune system, cell growth, adhesion, apoptosis, and angiogenesis. Until now 13 different types of galectins have been found in humans, among them Gal-1-4, 7-9 and 12 were detected in the normal endometrium. So far only Gal-1 and Gal-3 have been studied in relation to endometriosis. In a recent pilot study, the investigators have shown that Gal-9 levels are significantly elevated in the serum of endometriosis patients compared to healthy controls. Gal-9 had a high sensitivity (94%) and specificity (93,75%), indicating better diagnostic potential than that of other endometriosis biomarkers and of surgery as the current gold standard.

DETAILED DESCRIPTION:
Endometriosis is one of the most common infertility-related gynecologic disorder that affect approximately 10-15% of women in reproductive age. The main symptoms are chronic pelvic pain, infertility, dysmenorrhea and dyspareunia. The etiology and pathogenesis of endometriosis has been widely investigated over the past 30 years. Although there are several concepts trying to explain its development, but none of them can be applied for all types of the disease.

The peak incidence of the diagnosis of endometriosis lies between the ages of 25 to 34, although symptoms mostly develop much earlier. There exists an average diagnostic delay of 7 year but data widely varies between different countries: in the is UK 7.9 years, in the US 11.7 years, in Germany and Austria 7 years, in Spain 8 years, in Norway 6.7 years, in Ireland and Belgium 5 years and in Hungary 3.9 years. Such a diagnostic delay is multifactorial, but most importantly due to the lack of non-invasive diagnosis.

The current "gold standard" in the diagnosis of endometriosis remains a laparoscopy with a sensitivity of 79% and a specificity of 94%. Since laparoscopy is an invasive surgical procedure with its potential risk, the development of a non-invasive laboratory test would be of great benefit in the early, clinical management of this disease. Such a biomarker has the enormous potential to improve quality of life, reduce the risks to the patient and the enormous costs to society related to endometriosis.

Until now, several molecules involved in the pathogenesis of endometriosis were investigated as a potential biomarker, however the majority of them have proven inadequate for the diagnosis. In the past few years, lectins have become the focus of reproductive immunology, inflammation and autoimmunity. Galectins (Gal) are beta-galactoside binding lectins that play a key role in the regulation of the immune system, cell growth, adhesion, apoptosis, and angiogenesis. Until now 13 different types of galectins have been found in humans, among them Gal-1-4, 7-9 and 12 were detected in the normal endometrium. So far only Gal-1 and Gal-3 have been studied in relation to endometriosis. It was reported that Gal-1 had a cycle-dependent expression in normal endometrial stromal cells, and its production was significantly elevated in the early pregnancy decidua. In relation to endometriosis, Gal-1 was found to be more abundantly expressed in ectopic endometriotic lesions when compared with the eutopic tissues. Furthermore, the eutopic endometrium of the affected patients showed higher Gal-1 expression than its normal counterparts. In addition to this, similar to Gal-1, Gal-3 was overexpressed in various forms of endometriosis as well as in the eutopic endometrium of diseased women.

The investigators have previously shown that Gal-9 mRNA was markedly overexpressed in the eutopic endometrium of patients with endometriosis in comparison with healthy controls. In addition, the investigators results showed that besides the eutopic endometrium, Gal-9 was also expressed in ectopic implants regardless of the localization of the lesions. The investigators have determined that Gal-9 levels are significantly elevated in the serum of endometriosis patients compared to healthy controls. Gal-9 has a high sensitivity (94%) and specificity (93,75%), indicating better diagnostic potential than that of other endometriosis biomarkers. The optimal cutoff point estimated from the Youden's index was 132 pg/mL, with a sensitivity of 94% and specificity of 93.75%. Using this threshold, the positive predictive value was 97.92% and the negative predictive value was 83.33%, with a prevalence of 75.76%. The diagnostic accuracy of this test was 93.94%, indicating better diagnostic potential than that other already published serum biomarkers.

Based on this previous results, the investigators suggest that Gal-9 is produced by ectopic endometriotic implants, the investigators would like to determine the serum Gal-9 levels one day before and after the surgery and at least 1-6 months later. The investigators aim is to examine the serum Gal-1 and Gal-3 levels in endometriosis patients.

ELIGIBILITY:
Inclusion Criteria:

Histologically proved endometriosis

Exclusion Criteria:

Previous or current hormone therapy

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women in reproductive age
Study Population: in reproductive age laporoscopically proved endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Development of new non-invasive biomarker for endometriosis | 24 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brubel R, Bokor A, Pohl A, Schilli GK, Szereday L, Bacher-Szamuel R, Rigo J Jr, Polgar B. Serum galectin-9 as a noninvasive biomarker for the detection of endometriosis and pelvic pain or infertility-related gynecologic disorders. Fertil Steril. 2017 Dec;108(6):1016-1025.e2. doi: 10.1016/j.fertnstert.2017.09.008. PMID 29202955